CLINICAL TRIAL: NCT02589340
Title: Buspirone, in Combination With Amantadine, for the Treatment of Levodopa-induced Dyskinesia
Acronym: BUS-PD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathryn Anne Chung, Associate Professor - Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11875
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Parkinson's Disease; Dyskinesias; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Movement Disorders | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buspirone (Experimental): Two week titration up to 10 mg tablet/3 times a day for 7 days
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Two week titration up to 3 tablets/3 times a day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone
  Arms: Buspirone
Drug: Placebo — Sugar Pill
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of buspirone in combination with amantadine in reducing levodopa-induced dyskinesia (LID) in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Plan: We will perform a randomized, placebo-controlled, double-blind, two-period cross-over study to evaluate the safety, tolerability, and efficacy of a novel treatment combination for LID in PD.

Methods: Eligible subjects who consent to participate in this study will be randomized to one of two sequences of treatment interventions during the baseline visit. Each treatment sequence includes placebo and buspirone interventions. After randomization, each participant will titrate up on study drug for two weeks ending in 30 mg/day. At the end of each two week study drug period, the participant will then have a study visit at the VA Portland Health Care System that includes safety monitoring, adverse event monitoring, drug compliance, and several measurements of LID.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosis
* Currently taking a levodopa containing medication for Parkinson's disease
* Mild to Severe dyskinesia
* Currently taking between 200-500 mg of amantadine daily for treatment of levodopa-induced dyskinesia with insufficient suppression levodopa-induced dyskinesia.
* Stable medication regimen for at least 4 weeks prior to study.

Exclusion Criteria:

* Currently receiving any other treatment for levodopa-induced dyskinesia, including but not exclusive to deep brain stimulation.
* Not able to follow verbal commands
* Not able to stand unsupported for at least 60 seconds
* Not able to answer a patient questionnaire about their symptoms of Parkinson's disease and dyskinesia.
* Have proprioceptive deficits.
* Have a history of hepatic impairment
* Currently have severe renal impairment
* Currently have any other medical or psychiatric diagnosis that would preclude their ability to safely participate in the study.
* Significant cognitive impairment
* Pregnancy
* Breast-Feeding
* Unable to swallow study drug (capsule)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01; Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve - Dyskinesia - Forceplate | 6 hour levodopa dose cycle
  forceplate measurements of levodopa induced dyskinesia taken every 1/2 hour for 6 hours.
Dyskinesia - UDysRS | up to 6 weeks
  UDysRS total score comparison
Adverse Events | up to 6 weeks
  Adverse Events Monitoring/Frequency

CONTACTS AND LOCATIONS:
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS - DYSKINESIA. J Parkinsons Dis. 2019;9(3):449-465. doi: 10.3233/JPD-199002. No abstract available. PMID 31356217